CLINICAL TRIAL: NCT01393054
Title: Effect of Nigella Sativa Seed Extract on the Blood Pressure of Elderly With Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Aulia Rizka, MD, Faculty of Medicine University of Indonesia
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NS2602
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-07

CONDITIONS: Hypertension
Keywords: Nigella sativa seed extract; hypertension; elderly
MeSH Terms: conditions — Hypertension | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nigella sativa — Drug name: Nigella sativa seed extract in capsule Dosage 300 mg Frequency: twice daily Duration: 4 weeks

SUMMARY:
Despite of the development of new anti hypertensive agents, hypertension in elderly is still a big health problem. Nigella sativa seed extract, derived from a small plant originating in Middle east which can be found abundantly in Asia, has shown small antihypertensive effect in adult. Diuretic effect of Nigella sativa is thought to be the main mechanism for the effect but as it also shows anti-inflammatory and vasodilatory activity which are important contributors in arterial stiffness, the main pathogenesis of hypertension in elderly, thus it has a superior potential benefit for this population. We will conduct a randomized, double blind, placebo-controlled trial to prove the effect of Nigella sativa seed extract in elderly patients with hypertension. Our hypothesis is 300 mg Nigella sativa seed extract twice daily will have anti-hypertensive effect in the blood pressure of elderly with hypertension.

DETAILED DESCRIPTION:
The study will be conducted in Geriatric Outpatient Clinic of Cipto Mangunkusumo National Hospital, Jakarta, Indonesia.

Eligibility criteria are men and women over 60 years old and available to participate in the study for 4 weeks with blood pressure higher than 140/90.

Exclusion criteria are renal disease, hepatic failure, dementia and orthostatic hypotension and malignant hypertension.

Outcome measures are systolic and diastolic blood pressure after 4 weeks administration of 300 mg Nigella sativa seed extract twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Men and women more than 60 years old
* Systolic Blood Pressure 140 mm Hg AND OR diastolic blood pressure 90 mmHg
* Available during study duration (4 weeks)

Exclusion Criteria:

* Renal failure
* Hepatic failure
* Dementia
* Orthostatic hypotension
* Malignant hypertension

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure | 4 weeks
  We aim to measure the difference in systolic blood pressure after 4 weeks administration of 300 mg Nigella sativa seed extract in elderly with hypertension

SECONDARY OUTCOMES:
diastolic blood pressure | 4 weeks
  We measure the difference of diastolic blood pressure after 4 weeks administration of 300 mg Nigella sativa seed extract in elderly with hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Aulia Rizka, MD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (1):
- Cipto Mangunkusumo National Hospital, Jakarta, Jakarta Special Capital Region, Indonesia